CLINICAL TRIAL: NCT02664441
Title: Glucagon-Like Peptide-1 Agonist Effects on Energy Balance in Hypothalamic Obesity
Brief Title: Energy Balance & Weight Loss in Craniopharyngioma-related or Other Hypothalamic Tumors in Hypothalamic Obesity
Acronym: ECHO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Children's Hospitals and Clinics of Minnesota (Other); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Christian L Roth, MD, Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01DK104936-01A1 (NIH)
Record Dates: First submitted 2016-01-04; First posted 2016-01-27 (Estimated); Results first posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Hypothalamic Obesity
Keywords: Obesity; Drug intervention; Children; Adolescents; Young adults; Hypothalamic lesion; Change of weight status; Food intake; Energy expenditure; Hormonal changes; Glucagon-like peptide-1 agonist; Bydureon; Weight Loss; Energy balance
MeSH Terms: conditions — Sexual Infantilism; Obesity; Weight Loss | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide once weekly extended-release (Active Comparator): Injections of glucagon-like peptide (GLP)-1 agonist exenatide once weekly extended-release (Bydureon®) for 36 weeks in randomized intervention followed by 18 weeks open label exenatide once weekly extended-release.
  Interventions: Drug: Exenatide
- Matching placebo (Placebo Comparator): Weekly injections of placebo for 36 weeks followed by 18 weeks open label exenatide once weekly extended-release.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Exenatide — Weekly injections of active drug.
  Other Names: Bydureon®
  Arms: Exenatide once weekly extended-release
Drug: placebo — Weekly placebo injections
  Arms: Matching placebo

SUMMARY:
The proposed multicenter study will test the effect of glucagon-like peptide (GLP)-1 agonist exenatide once weekly extended-release (ExQW, Bydureon®) on clinical outcomes and metabolic parameters in a double-blind, placebo-controlled 36 week randomized trial with an 18 week open label extension. Following baseline testing, 48 patients will be randomly assigned with equal allocation to ExQW or matching placebo injection for 36 weeks, followed by an 18 week open label extension during which all patients receive ExQW. Changes of weight status, body composition, free-living total daily energy expenditure (EE) by doubly labeled water (DLW), activity by acetimetry, energy intake (questionnaires and food diary), as well as glucose tolerance and hormonal parameters of energy homeostasis and insulin resistance will be assessed before treatment and at the end of the placebo-controlled phase (week 36). Activity, metabolic outcomes, energy intake will be also assessed at study week 18 (mid treatment of randomized study), as well as week 54 (end of open label treatment).

DETAILED DESCRIPTION:
Excessive weight gain and its cardiometabolic sequela are frequent complications of hypothalamic tumors, a condition known as hypothalamic obesity (HO). Most tumors in this region are craniopharyngiomas (CP),1 which constitute 5-9% of childhood brain tumors. Patients with CP typically become obese and have more features of the metabolic syndrome compared to matched controls. Overall, a 3-19-fold higher cardiovascular mortality had been reported, and a recent nationwide population-based study in Sweden demonstrated increased rates for cerebral infarction (7-fold), death due to cerebrovascular diseases (5-fold), and type 2 diabetes mellitus (6-fold) in CP patients in comparison to the general population. Thus, early and effective management of obesity is vital for this population, which is more resistant to treatment than uncomplicated obesity. Recognized risk factors for severe obesity include large hypothalamic tumors or lesions affecting several medial and posterior hypothalamic nuclei that impact satiety signaling pathways. Structural damage in these nuclei often lead to uncontrolled appetite, rapid weight gain, central insulin and leptin resistance, decreased sympathetic activity, low energy expenditure (EE), and increased energy storage in adipose tissue. Recently, the investigators developed a semi-quantitative assessment of hypothalamic damage on brain magnetic resonance imaging (MRI) to predict the risk for HO development in CP.

Previous results of treating HO with a glucagon-like-peptide-1 receptor agonist (GLP1RA) in rats and humans provide promising proof-of-principle data to support this current randomized clinical trial. The primary hypothesis of this study is that drugs causing weight loss via intact hindbrain signaling pathways offer a desperately needed option for treatment of HO, even in very obese HO subjects with severe hypothalamic damage. Induction of weight loss by GLP1RAs is believed to be related to multiple mechanisms involving the gastrointestinal tract, vagus nerve, and the brain leading to increased satiety. Peripheral administration of GLP-1 or GLP1RA reduces blood glucose and energy intake in humans and rodents, and long-term treatment results in loss of body weight. Critically, the investigators do not know whether GLP1RA treatment affects EE and activity, or whether the site and size of brain lesions affect responses to GLP1RA treatment.

The investigators' previous clinical studies of the GLP1RA exenatide in obese adolescents and adults have generated the critical safety and efficacy data needed to design a clinical trial. In a pilot study conducted at Children's Hospitals and Clinics of MN, pretreatment hyperphagia was associated with BMI reduction. Using these data, the investigators have designed a prospective, multicenter trial that will examine the effects of GLP1RA on BMI, cardiovascular disease (CVD) risk factors, energy homeostasis and other factors in subjects with HO secondary to CP.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-25 years at time of enrollment
* Diagnosis of hypothalamic obesity with age- and sex adjusted BMI ≥ 95% or BMI ≥30 kg/m² if over 18 y
* History of craniopharyngioma or another tumor located in the hypothalamic area
* Hypothalamic lesion documented by neuroradiology
* ≥ 6 months post-surgical or radiation treatment
* Weight stable or increasing over 3 months prior to screening visit
* Stable hormone replacement for at least 3 months prior to screening visit

Exclusion Criteria:

* Renal impairment (GFR<60 ml/min/1.73m² using the Schwarz formula)
* History of gastroparesis; pancreatitis or gallstones (unless status post cholecystectomy)
* Family history of multiple endocrine neoplasia type 2 or familial medullary thyroid carcinoma metabolic disorders
* Any insulin-treated diabetes mellitus, poorly controlled type 2 diabetes (HbA1c ≥ 10%), or any other chronic serious medical conditions such as cardiovascular disease, malignancy or hematologic disorder, complicated syndromic disorder, or psychiatric disorders (schizophrenia, major depression, history of suicide attempts)
* Calcitonin >50 mg/L at screening
* Initiation of weight loss medications within 3 months of screening visit
* Previous donation of blood >10% of estimated blood volume within 3 months prior study
* Current warfarin use
* Current use of any other GLP1 receptor agonist
* Untreated thyroid disorder or adrenal insufficiency
* History of bariatric surgery or planned bariatric surgery until end of study
* Pregnancy, lactation or expectation to conceive during study period
* Subject unlikely to adhere to study procedures in opinion of investigator
* Subject with contraindication to neuroimaging by MRI

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2016-03; Primary Completion 2020-03-16 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Roth, MD, Principal Investigator — Seattle Childrens
Locations (3):
- United States (3):
  - Children's Hospitals adn Clinics of Minnesota, Minneapolis, Minnesota
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Seattle Childrens, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients aged 10-25 years of age with a diagnosis of hypothalamic obesity following treatment for craniopharyngioma were recruited from pediatric endocrinology outpatient clinics at the three research sites (Seattle Children's Hospital, Seattle, WA, USA; Children's Minnesota, St. Paul, MN, USA; and Vanderbilt University Medical Center, Nashville, TN, USA) and hypothalamic obesity internet support groups.
Pre-assignment Details: Qualified participants started with a 2-week placebo run-in to test adherence to the protocol prior to randomization.
Period: Randomization
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Started | 23 | 19
Completed | 23 | 18
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: 36-week Randomized Trial
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Started | 23 | 18
Completed | 20 | 15
Not Completed | 3 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3
Period: 18-week Open Label Extension
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Started | 20 | 15
Completed | 17 | 14
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Categorical [Count of Participants; unit: Participants] — Population: One participant withdrawn in placebo group
  Participants
    <=18 years | 16 | 14 | 30
    Between 18 and 65 years | 7 | 5 | 12
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Years as continuous measure
  years | 16.9 (4.3) | 16.9 (4.7) | 16.9 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 21 | 19 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 21 | 16 | 37
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 19 | 42
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] — Calculated by the formula: body weight in kg divided by height in meters².
  kg/m² | 35.8 (6.6) | 38.7 (7.5) | 37.3 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Body Mass Index (BMI) as Calculated by the Formula: Body Weight in kg Divided by Height in Meters².
Description: Percent change of body mass index (BMI), as calculated by the formula: body weight in kg divided by height in meters², between baseline and the end of the 36-week randomized drug treatment phase.
Time Frame: From baseline to 36 weeks
Population: Analyses include all participants randomized to a study drug and received at least one drug treatment administration. Missing data was imputed using a last observation carry-forward approach.
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Number analyzed (Participants) | 23 | 18
percent change from baseline | 1.7 (0.8) | 3.5 (0.9)
Statistical Analysis 1: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Test type: Superiority; p = 0.40, Mixed Models Analysis; Randomization stratification variables (site, sex and age group) were used as covariates; Mean Difference (Net) = -1.7, 95% CI 2-sided [-4.1 to 0.6]

2. Secondary Outcome: Changes in Body Composition as Assessed by Body Fat Mass Using Dual Energy X-ray Absorptiometry (DEXA)
Description: Body composition change between baseline and the end of the 36-week randomized drug treatment phase assessed by dual energy x-ray absorptiometry (DEXA) and expressed as the change in adipose tissue mass.
Time Frame: At baseline and 36 weeks
Population: Of the 41 enrolled participants, 20 out of 23 participants randomized to exenatide once weekly extended-release and 15 out of 18 participants randomized to placebo completed both pre- and post-treatment assessments and are included in this analysis.
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Number analyzed (Participants) | 20 | 15
kilograms | 1.5 (0.9) | 4.6 (1.0)
Statistical Analysis 1: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Test type: Superiority; p = 0.02, Mixed Models Analysis; Randomization stratification variables (site, sex and age group) were used as covariates; Mean Difference (Net) = -3.1, 95% CI 2-sided [-5.7 to -0.4]

3. Secondary Outcome: Changes in Fat and Total Calorie Intake Assessed by Free Buffet Meal Analysis.
Description: Changes in fat and total calorie intake during free buffet meals assessed at baseline and after 36-weeks of study drug treatment.
  The buffet meal is an objective measure of satiety as it assesses food intake and choice after a caloric preload. A standardized test meal preload provided 20% of estimated daily caloric requirements,based on the Schofield-HW equation. The purpose of the test meal is to ensure that study participants are in an equally fed state. Ninety minutes later, an ad libitum buffet meal was served consisting of a wide variety of food items and more than the child's estimated daily calorie requirements will be offered (5,000 kcal). Children had access to the buffet for 30 min, after which calorie intake and composition of consumed foods was measured by weighing back uneaten food.
Time Frame: From baseline to 36 weeks
Population: Of the 41 enrolled participants, 18 out of 23 participants randomized to exenatide once weekly extended-release and 15 out of 18 participants randomized to placebo completed both pre- and post-treatment assessments and are included in this analysis.
Measure: Mean (Standard Error); unit: grams
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Number analyzed (Participants) | 18 | 15
grams
  Fat Intake | -9.5 (6.3) | 14.5 (7.7)
  Total Calorie Intake | -287 (130) | 224 (136)
Statistical Analysis 1: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Analysis for Fat Intake; Test type: Superiority; p = .032, Regression, Linear; Adjusted for baseline values; Mean Difference (Final Values) = -20.2, 95% CI 2-sided [-37.8 to -2.7]
Statistical Analysis 2: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Analysis for Total Calorie Intake; Test type: Superiority; p = .02, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = -430, 95% CI 2-sided [-761 to -100]

4. Secondary Outcome: Changes in Fasting Glucose
Description: Change in fasting blood glucose between baseline and the end of the 36-week randomized drug treatment phase.
Time Frame: From baseline to 36 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Number analyzed (Participants) | 23 | 18
mg/dL | 7.4 (6.0) | 3.7 (3.5)
Statistical Analysis 1: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Test type: Superiority; p = 0.19, Mixed Models Analysis; Randomization stratification variables (site, sex and age group) as covariates; Geometric Mean Ratio = 1.42, 95% CI 2-sided [0.97 to 2.08] — Data were log-transformed prior to analysis. Results were back-transformed through exponentiation and presented as geometric mean ratios with 95% confidence intervals

5. Secondary Outcome: Changes in HDL Cholesterol and Triglycerides Assessed by Fasting Lipids
Description: Change in fasting HDL cholesterol and triglycerides between baseline and the end of the 36-week randomized drug treatment phase.
Time Frame: From baseline to 36 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Number analyzed (Participants) | 23 | 18
mg/dL
  HDL Cholesterol | 0.7 (2.1) | 0.6 (2.8)
  Triglycerides | -0.6 (8.1) | 4.2 (8.6)
Statistical Analysis 1: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Analysis for HDL Cholesterol; Test type: Superiority; p = 0.82, Mixed Models Analysis; Randomization stratification variables (site, sex and age group) as covariates; Geometric Mean Ratio = 1.00, 95% CI 2-sided [0.91 to 1.11] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Analysis for Triglycerides; Test type: Superiority; p = 0.92, Mixed Models Analysis; Randomization stratification variables (site, sex and age group) as covariates; Geometric Mean Ratio = 1.00, 95% CI 2-sided [0.83 to 1.19] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Changes in Inflammation Assessed by C-reactive Protein (CRP)
Description: Change in C-reactive protein (CRP) between baseline and the end of the 36-week randomized drug treatment phase.
Time Frame: From baseline to 36 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Number analyzed (Participants) | 23 | 18
mg/dL | 0.00 (0.07) | 0.18 (0.27)
Statistical Analysis 1: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Test type: Superiority; p = 0.03, Mixed Models Analysis; Randomization stratification variables (site, sex and age group) as covariates; Geometric Mean Ratio = 0.62, 95% CI 2-sided [0.41 to 0.92] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Changes of Insulin Resistance Assessed by Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: Changes of insulin resistance estimated by the homeostasis model assessment of insulin resistance (HOMA-IR) using the formula HOMA-IR = insulin [mU/l] x glucose [mmol/l]) / 22.5 where both insulin and glucose values are obtained from a fasting blood sample.
Time Frame: From baseline to 36 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: HOMA-IR score
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Number analyzed (Participants) | 23 | 17
HOMA-IR score | 3.5 (1.7) | 2.2 (2.4)
Statistical Analysis 1: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Test type: Superiority; p = 0.32, Mixed Models Analysis; Randomization stratification variables (site, sex and age group) as covariates; Geometric Mean Ratio = 1.39, 95% CI 2-sided [0.90 to 2.14] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: Changes of Circulating Leptin Levels
Description: Change in circulating leptin between baseline and the end of the 36-week randomized drug treatment phase.
Time Frame: From baseline to 36 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Number analyzed (Participants) | 23 | 18
ng/mL | 1.4 (6.3) | 11.8 (9.4)
Statistical Analysis 1: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Test type: Superiority; p = 0.69, Mixed Models Analysis; Randomization stratification variables (site, sex and age group) were used as covariates; Geometric Mean Ratio = 0.95, 95% CI 2-sided [0.81 to 1.10] — [estimate comment as in outcome 4, analysis 1]

9. Secondary Outcome: Changes of Energy Expenditure Assessed by Doubly Labeled Water Analysis
Description: Total energy expenditure in the free-living environment was measured using doubly labeled water which estimates carbon dioxide production by measuring the elimination of the tracers deuterium (²H) and oxygen-18 (¹⁸O) from the body. These measures are used to determine the average daily rate of carbon dioxide production which is then used to calculate total energy expenditure using an equation from Weir and an assumed food quotient (0.85).
Time Frame: Baseline and 36 weeks
Population: Of the 41 enrolled participants, 19 out of 23 participants randomized to exenatide once weekly extended-release and 14 out of 18 participants randomized to placebo completed both pre- and post-treatment assessments and are included in this analysis.
Measure: Mean (Standard Error); unit: kcals/day
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Number analyzed (Participants) | 19 | 14
kcals/day | -17.8 (38.0) | 146.3 (29.0)
Statistical Analysis 1: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Test type: Superiority; p = 0.004, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = -166.4, 95% CI 2-sided [-269.7 to -63.1]

10. Secondary Outcome: Changes of Energy Intake Assessed by Automated Self-Administered 24-Hour Dietary Recall (ASA24-Kids)
Description: Self-reported daily energy intake was assessed by Automated Self-Administered 24-Hour Dietary Recall (ASA24-Kids, http://appliedresearch.cancer.gov/tools/instruments/asa24/), a web-based diet assessment tool that allows 24-hour diet recall using branded food items.
Time Frame: Baseline and 36 weeks
Population: Of the 41 enrolled participants, 14 out of 23 participants randomized to exenatide once weekly extended-release and 9 out of 18 participants randomized to placebo completed both pre- and post-treatment assessments and are included in this analysis.
Measure: Mean (Standard Error); unit: kcals
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Number analyzed (Participants) | 14 | 9
kcals | -62 (155) | -210 (336)
Statistical Analysis 1: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Test type: Superiority; p = 0.58, Regression, Linear; Adjusted for baseline; Mean Difference (Net) = -145.0, 95% CI 2-sided [-653.5 to 363.4]

11. Secondary Outcome: Changes in Glucose 120 Minutes Following an Oral Glucose Tolerance Test
Description: Change in blood glucose measures 120 minutes post-glucose bolus during an oral glucose tolerance test between baseline and the end of the 36-week randomized drug treatment phase.
Time Frame: From baseline to 36 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly Extended-release | Matching Placebo
Number analyzed (Participants) | 23 | 18
mg/dL | -12.4 (10.9) | -3.4 (3.7)
Statistical Analysis 1: Comparison: Exenatide Once Weekly Extended-release vs Matching Placebo; Test type: Superiority; p = 0.088, Mixed Models Analysis; Randomization stratification variables (site, sex and age group) were used as covariates; Mean Difference (Net) = -8.5, 95% CI 2-sided [-19.1 to 2.1]

ADVERSE EVENTS:
Time Frame: Double-Blind Randomized Phase - From Study Visit 1 (0 weeks) through end of Study Visit 4 (36 weeks); Open Label Extension - From Study Visit 4 (36 Weeks) through end of Study Visit 5 (54 weeks)
Groups:
- Double-Blind Exenatide Once Weekly Extended-release: Injections of glucagon-like peptide (GLP)-1 agonist exenatide once weekly extended-release (Bydureon®) for 36 weeks in randomized intervention
  Exenatide: Weekly injections of active drug.
- Double-Blind Placebo: Weekly injections of placebo for 36 weeks in randomized intervention
  placebo: Weekly placebo injections
- Open Label Exenatide Once Weekly Extended-release: 18 weeks open label exenatide once weekly extended-release (Bydureon®) arm.
  Exenatide: Weekly injections of active drug.
Arm/Group | Double-Blind Exenatide Once Weekly Extended-release | Double-Blind Placebo | Open Label Exenatide Once Weekly Extended-release
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/18 | 1/35
Serious Adverse Events (participants affected / at risk) | 2/23 | 1/18 | 4/35
Other Adverse Events (participants affected / at risk) | 21/23 | 15/18 | 17/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Exenatide Once Weekly Extended-release (N=23) | Double-Blind Placebo (N=18) | Open Label Exenatide Once Weekly Extended-release (N=35)
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cholecystitis / Cholecystectomy (Hepatobiliary disorders) | 0 | 0 | 1
Hypernatremic dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Migraine Headache (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1
Altered mental status (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Exenatide Once Weekly Extended-release (N=23) | Double-Blind Placebo (N=18) | Open Label Exenatide Once Weekly Extended-release (N=35)
Abdominal pain (Gastrointestinal disorders) | 9 | 2 | 1
Nausea (Gastrointestinal disorders) | 6 | 3 | 3
Diarrhea (Gastrointestinal disorders) | 7 | 3 | 4
Vomiting (Gastrointestinal disorders) | 4 | 4 | 5
Constipation (Gastrointestinal disorders) | 3 | 2 | 2
Cholelithiasis (Gastrointestinal disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 2
Headache (Nervous system disorders) | 7 | 6 | 3
Injection site reaction (General disorders) | 7 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT02664441/Prot_SAP_000.pdf